CLINICAL TRIAL: NCT00678522
Title: The Acute Effect of Atorvastatin on Renal Sodium Excretion, Glomerular Filtration Rate, Tubular Function and Vasoactive Hormones in Patients With Non-Insulin Dependent Type II Diabetes.
Brief Title: The Acute Effect of Atorvastain on Renal Function in Patients With Type II Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Regional Hospital Holstebro (Other)
Collaborators: Medical Research (Ambiguous)
Responsible Party: Lone Paulsen, Medical Research
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: MED.RES.HOS.2006.04.LP
Record Dates: First submitted 2008-05-13; First posted 2008-05-15 (Estimated); Last update posted 2008-05-15 (Estimated); Status verified 2008-05

CONDITIONS: Healthy Subjects
Keywords: Atorvastatin; Renal function; Hemodynamics; Diabetes type II; sodium excretion
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Atorvastatin — 80 mg atorvastatin daily on two following days

SUMMARY:
We wanted to test the hypothesis that acute treatment with atorvastatin changes renal sodium excretion, glomerular filtration rate, tubular function and vasoactive hormones in patients with type II diabetes, not in treatment with insulin.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 40-70 yrs
2. estimated GFR between 30 and 90 ml/min
3. BMI<35
4. Fertile women had to use oral contraceptives or IUD
5. HbA1c< 10%
6. Urine-albumin<1,5 g/l

Exclusion Criteria:

1. Treatment with insulin
2. Cerobrovascular insult or other disease of the brain
3. Insufficiency of the heart or lungs
4. Liverdisease with ALAT > 200 U/L
5. hemoglobin < 7,0 mmol/l
6. Cancer
7. Alcohol abuse
8. Medical treatment with psycopharmaca or/and analgetics
9. Pregnancy and breast feeding, 10 blood donation one month before the study.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2007-09; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
GFR, clearance of sodium and lithium, fractional excretion of sodium and lithium, U-AQP-2, total sodium excretion, albumin excretion rate and free water clearance. | 6 months

SECONDARY OUTCOMES:
AVP, Ang-II, Aldo, ANP, BNP, PRC, BP, HR. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Erling B. Pedersen, Professor, Principal Investigator — Dept. of medical reaserch, Holstebro Hospital, Denmark
Locations (2):
- Denmark (2):
  - Medical Reseach, Holstebro Hospital, Holstebro
  - Department of Medical Research, Holstebro Hospital, Holstebro